CLINICAL TRIAL: NCT03309345
Title: - Contribution of Diet Induced Thermogenesis (DIT) and Fat Oxidation to Body Fatness and Body Composition of Patients With Phenylketonuria - Contribution of Physical Activity Energy Expenditure and Energy Intake to Body Fatness and Body Composition of Patients With Phenylketonuria
Brief Title: Body Composition, Energy Intake and Expenditure in People With Phenylketonuria
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Konstantinos Gerasimidis, Lecturer in Clinical Nutrition, University of Glasgow
Other Study IDs: R&D:GN16ME448P, REC:16/SW/0288
Record Dates: First submitted 2017-06-23; First posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Phenylketonuria (PKU)
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group, PKU group: Children and adults (10 - 45 years old) with PKU attending the metabolic medicine clinics in the area of National Health Services (NHS) Greater Glasgow and Clyde (GGC) will be approached for recruitment. Participants will be free from history of acute and chronic illness (other than PKU) requiring regular appointments to the doctor and/or chronic use of medication or major gastrointestinal surgery where major part of the gut has been resected as these conditions are known to impact on energy expenditure and dietary intake. Pregnant or lactating women will also be excluded from participation. People with learning or mobility difficulties or those with incapacity to provide informed consent will be excluded too. The clinical treatment team will evaluate patients' capacity to consent before considering them to participate in the study.
  Interventions: Other: No intervention
- Control group, healthy control: Gender, BMI and age matched healthy people will be recruited as a control group. Pregnant or lactating women will be excluded from participation. Those with any chronic illnesses or bone injuries will also be excluded.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention as this is an observational study investigates the difference between PKU ant matched healthy control in terms of energy components and dietary intake

SUMMARY:
This will be case-control study investigating whether dietary intake and components of energy expenditure such as Basal metabolic rate (BMR), physical activity energy expenditure (PAEE) and diet induce thermogenesis (DIT) are different between people with phenylketonuria (PKU) and matched healthy controls. Participants will be children and adults with PKU age between 10 to 45 years old, free from history of any acute and chronic illness. Participants will attend the Metabolic Research Unit at New Lister Building (NLB) after 12-hour overnight fasting refraining from alcohol consumption for at least 24 hours. Any planned exercise will be avoided during the 48 hours prior visit to the Metabolic Research Unit. Height, body weight and handgrip strength will be measured upon arrival at the unit. BMR will be assessed and participants will be asked to provide baseline saliva sample followed by consumption of 8 g deuterium water (D2O) diluted in drinking water. Normal or PKU-type isocaloric breakfast meal will then be provided based on intervention group-type. DIT will be measured 5 times for 3 hours, with each measurement lasting for 20 minutes. Two saliva samples will be collected at 3 and 3.5 hours after ingestion of D2O. Participants will be asked to perform an incremental intensity exercise test for 20 minutes on the treadmill during which expired air will be collected and accelerometer counts and heart rate will be measured. Participants will then be trained on how to recorded food intake and how to use accelerometers for habitual physical activity measurements. PKU participants (and their parents if ≤15 years old) will be asked to complete quality of life (QoL) questionnaires. Participants will be required to wear the accelerometer equipment for seven consecutive days excluding bedtime and keep a record of non-wear times. During these days, they will also prospectively record estimated food and beverages intake over four days including one weekend day.

DETAILED DESCRIPTION:
1. Anthropometric measurements:

   Height will be measured using a wall-mounted stadiometer to the nearest 0.01 meter. Body mass will be measured in kilograms using balance scale. Body mass index (BMI) will be calculated using the following formula: BMI = kg/m² [weight in kilograms/ height in meters²].
2. Handgrip strength (kilograms):

   Grip strength will be measured by using a handgrip dynamometer as a measure of strength and physical capacity.
3. Body composition determination, saliva samples collection, storage and analysis:

   Body composition will be determined using the deuterium water (D2O) dilution technique. Participants will be provided a dose of 8 g of D2O diluted in drinking water. Participants will be asked to provide a baseline saliva samples and another samples will be obtained at 3 and 3.5 hrs after ingestion of the D2O. Samples will be stored in freezers at -20 °C. All samples will be analysed at Scottish Universities Environmental Research Centre (SUERC), Glasgow, for measurements of total body water (TBW) by means of Fourier Transform Infrared Spectrometry (FTIR).
4. Metabolic rate measurement:

   Metabolic rate will be measured by means of computerised open-circuit ventilated hood system (Quark, Resting metabolic rate (RMR) ®, Italy). Rate of oxygen consumption (O2) and carbon dioxide production (CO2) will be recorded every 30 seconds for total duration of 20 minutes with 10 minute break.
5. Breakfast meal:

   Participants in phenylketonuria (PKU) group will receive a breakfast based on PKU-type foods. Participants in control group will receive a similar breakfast based on normal foods with calories content and weight being matched between the groups.
6. Measurements of physical activity (PA) and physical activity energy expenditure (PAEE):

   ActiGraph accelerometer (GT3X+®) will be used to measure and record acceleration of participant's physical activity. The participants will have to wear them for seven consecutive days. They should record the time they put the monitor on in the morning and when taking it off in the evening in their activity diaries. They also have to keep notes of time and reason if they take the monitor off during the day.

   Individual calibration curves for counts against rate of O2 and rate of CO2 will be established during rest, and continuous incremental exercise test on the treadmill. Each participant will conduct walking/ running test with starting speed of 2 km/h being increased by 1 km/h every 4 minutes. The test will be stopped when heart rate (HR) just reaches 80 % of maximal heart rate (HRmax) defined as 220 - age. During this incremental test, participants will wear both ActiGraph accelerometer and face mask connected to indirect calorimetry equipment (Quark RMR®, Italy) to measure rate of O2 and rate of CO2.
7. Dietary analyses:

   Participants will record their food intake by food portion size estimation method. Participants will be asked to record their intake for four days including one weekend day. Data from food diaries will be compared to reference UK photographic atlas of food portion sizes to estimate weight of food intake. Food and energy intake will then be calculated using computerised program.
8. Quality of life assessment:

   PKU participants' quality of life will be assessed by means of validated PKU-specific Health-related Quality of Life Questionnaires (PKU-QOL). The questionnaires cover the physical, emotional, and social impacts of PKU and its treatment on patients' lives and come along with a software to calculate PKU-QoL scores.
9. Clinical data on history of disease activity:

Information about disease management relevant to the study (i.e. records of phenylalanine levels, weight and height status, and number of protein exchanges and dietary compliance, quantity and types of prescribed PKU foods and amino acid supplements) will be collected from the patients' medical notes. The data will be obtained for one year prior to the participants' intended day of study start.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults with PKU between 10 to 45 years old
* Free from history of any acute and chronic illness (other than PKU)

Exclusion Criteria:

* Patients with learning or mobility disabilities
* Patients who are deemed not competent to provide informed consent as judged by the clinical staff
* Pregnant or lactating women
* Participants who are not able to read, comprehend or communicate in English

Ages: 10 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Eligible patients will be identified from the clinical appointment lists held by the medical team of the metabolic medicine clinics in NHS GGC. A member of the treatment team (Mrs Barbara Cochrane or other members of the primary management clinical teams) will send an introductory letter about the study and the study information leaflet to those participants who are eligible to participate. This will give adequate time for the participants and their carers to consider the study prior to their subsequent clinical appointment. To increase recruitment rate, the researchers will present the study at the PKU group sessions, cooking and social events that are organised by the local clinical team
  Controls will be recruited by means of poster advertisement and by university's email-broadcasting and word of mouth in the campus of the University of Glasgow, and other public areas (libraries, train/bus stations).
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-01-20 (Estimated); Study Completion 2019-01-20 (Estimated)

PRIMARY OUTCOMES:
Basal metabolic rate (BMR) | 14 months
  BMR by means of computerised open-circuit ventilated hood system (Quark RMR®, Italy).
Diet induce thermogenesis (DIT) | 14 months
  DIT will be measured by means of computerised open-circuit ventilated hood system (Quark RMR®, Italy).
Physical activity energy expenditure (PAEE) | 14 months
  PAEE will be calculated during rest, and continuous incremental exercise by establishing an individual calibration curves for counts accelerometer against rate of oxygen (O2) and rate of carbon dioxide (CO2).
Energy and macro-nutrient intake | 14 months
  Participants will be asked to estimate their food intake using household measures or natural unit sizes (e.g. slices of bread) and to record their intake for four days including one weekend day.
  Data from food diaries will be compared to reference UK photographic atlas of food portion sizes to estimate weight of food intake. Food and energy intake will then be calculated using the dietary software 2010 (The Robert Gordon University, Aberdeen, Scotland, UK).

SECONDARY OUTCOMES:
Body composition | 14 months
  Will be determined using the deuterium water (D2O) dilution technique
Quality of life assessment | 14 months
  PKU participants' quality of life will be assessed by means of validated PKU-specific Health related Quality of Life Questionnaires (PKU-QOL)
Hand-grip strength | 14 months
  Grip strength will be measured by using a hand-grip dynamometer as a measure of strength and physical capacity

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Malkova, BSc,MSc,PhD, Study Director — University of Glasgow; Konstantinos Gerasimidis, PhD,MSc,APHNutr, Principal Investigator — University of Glasgow; Barbara Cochrane, BSc,MSc, Study Director — Queen Elizabeth University Hospital; Sarah Adam, BSc,PGC, Study Director — Glasgow Royal Infirmary Hospital; Peter Galloway, Med,MB CHB,DCH,FRCP,FRCPath, Study Director — Glasgow Royal Infirmary Hospital
Locations (1):
- University of Glasgow, Glasgow, Scotland, United Kingdom